CLINICAL TRIAL: NCT07133763
Title: A Multicenter, Single-Arm, Prospective Study to Evaluate the Efficacy and Safety of PD-1 Inhibitor Combined With Tenofovir, Chidamide, and Lenalidomide in the Treatment of Relapsed or Refractory EBV-Associated Lymphoproliferative Disorders.
Brief Title: Application of PD-1 Inhibitors, Tenofovir, Chidamide, and Lenalidomide in Relapsed/Refractory EBV-associated Lymphoproliferative Disorders.
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Affiliated Hospital of Xuzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XYFY2025-KL293-01
Record Dates: First submitted 2025-08-04; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: EBV-Associated Lymphoproliferative Disorders; PD-1 Inhibitor; Tenofovir; Chidamide; Lenalidomide
Keywords: EBV-Associated Lymphoproliferative Disorders; PD-1 Inhibitor; tenofovir; Chidamide; lenalidomide
MeSH Terms: interventions — Tenofovir; N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Evaluate efficacy and safety of multi-drug therapy in EBV-Associated Lymphoproliferative Disorders. (Experimental): To investigate the therapeutic effect of PD-1 inhibitor combined with tenofovir, chidamide, and lenalidomide in EBV-Associated Lymphoproliferative Disorders, and to evaluate its safety and clinical benefit in this patient population.
  Interventions: Drug: PD-1 Inhibitor Combined with Tenofovir, Chidamide, and Lenalidomide for the Treatment of EBV-Associated Lymphoproliferative Disorders.

INTERVENTIONS:
Drug: PD-1 Inhibitor Combined with Tenofovir, Chidamide, and Lenalidomide for the Treatment of EBV-Associated Lymphoproliferative Disorders. — This study investigates a novel multi-targeted regimen combining a PD-1 inhibitor, tenofovir, chidamide, and lenalidomide for relapsed/refractory EBV-associated lymphoproliferative disorders (LPDs). Unlike conventional therapies focused on antivirals or chemotherapy alone, this approach integrates antiviral suppression, epigenetic reactivation, immune modulation, and checkpoint blockade to achieve synergistic antitumor and antiviral effects. Preliminary data show effective EBV inhibition and tumor regression. This strategy offers a promising and distinct therapeutic option for EBV-driven lymphoid malignancies resistant to standard treatment.

SUMMARY:
This study is a prospective, multicenter, single-arm clinical trial designed to evaluate the efficacy and safety of PD-1 inhibitor combined with tenofovir, chidamide, and lenalidomide in the treatment of relapsed or refractory Epstein-Barr virus (EBV)-associated lymphoproliferative disorders (LPDs). The primary endpoint is the overall response rate (ORR) at 3 months, including complete response (CR) and partial response (PR). Secondary endpoints include overall survival (OS), progression-free survival (PFS), as well as safety and tolerability assessments. Eligible patients must have histologically confirmed EBV-positive B-cell or T/NK-cell LPDs with measurable lesions. This combination regimen targets multiple mechanisms, including inhibition of EBV replication, activation of the immune system, and enhancement of antitumor effects, aiming to provide an innovative therapeutic strategy for this challenging disease.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed EBV-associated lymphoproliferative disorders, including EBV-positive B-cell LPD and EBV-positive T/NK-cell LPD, with EBV-encoded RNA (EBER)+ by in situ hybridization, or EBV nuclear antigen (EBNA)+, or latent membrane protein (LMP1/2)+ in the lesion tissue.
2. Age ≤75 years with an ECOG performance status ≤2.
3. At least one bidimensionally measurable lesion for evaluation: for nodal lesions, longest diameter ≥1.5 cm and shortest diameter ≥1.0 cm; for extranodal lesions, longest diameter ≥1.0 cm; or ≥20% monoclonal EBV-infected lymphocytes detected by flow cytometry.
4. Expected survival of more than 3 months.
5. Ability to comply with follow-up. Patients must be aware of the nature of their disease and voluntarily agree to participate in the study and follow-up.

Exclusion Criteria:

1. Patients with impaired liver or kidney function, defined as serum direct bilirubin, indirect bilirubin, and/or ALT, AST, or serum creatinine levels >2 times the upper limit of normal, unless deemed lymphoma-related.
2. Patients with bone marrow failure, defined as absolute neutrophil count (ANC) <1.5×10⁹/L or platelets <75×10⁹/L, unless the hematologic abnormalities are considered due to bone marrow infiltration by lymphoma.
3. Patients who have experienced grade ≥3 neurotoxicity within the past 2 weeks.
4. Patients with chronic heart failure classified as NYHA Class III or IV, or with left ventricular ejection fraction <50%, or with a history within the past 6 months of any of the following: acute coronary syndrome, acute heart failure (Class III or IV), or significant ventricular arrhythmias (e.g., sustained ventricular tachycardia, ventricular fibrillation, or post-resuscitation sudden cardiac arrest).
5. Patients with AIDS, syphilis, or active hepatitis B (HBV DNA >1×10⁴ copies/ml) or active hepatitis C infection.
6. Patients diagnosed with malignancies other than lymphoma or currently undergoing treatment for other cancers, except:

   ① Those who have received curative treatment and have been disease-free for ≥5 years prior to enrollment;

   ② Patients with adequately treated, non-melanoma skin cancers such as basal cell carcinoma without evidence of disease;

   ③ Patients with adequately treated carcinoma in situ of the cervix without evidence of disease.
7. Patients with other hematologic diseases (e.g., hemophilia, myelofibrosis) considered unsuitable for the study by the investigator.
8. Patients with severe active infections.
9. Patients who underwent Grade 2 or higher surgery within 3 weeks before treatment initiation.
10. Patients with a history of substance abuse, or medical, psychological, or social conditions that may interfere with study participation or evaluation, as judged by the investigator.
11. Any other condition the investigator considers unsuitable for study enrollment.
12. Known hypersensitivity to any component of the investigational drugs.

Ages: 0 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the 3-month overall response rate (ORR), including complete and partial responses, in relapsed/refractory EBV-associated LPD patients treated with PD-1 inhibitor, tenofovir, chidamide, and lenalidomide. | After 3 months of treatment according to the study protocol, a comprehensive efficacy assessment will be conducted. Patients achieving CR or PR will continue treatment, while those with SD or PD will be withdrawn from the study.

SECONDARY OUTCOMES:
24-month Overall Survival Rate in Relapsed/Refractory EBV-Associated Lymphoproliferative Disorders. | From first dose until death from any cause (assessed at 24 months）
  Proportion of patients alive at 24 months after initiation of tirelizumab combination therapy.
24-month Progression-free Survival Rate in Relapsed/Refractory EBV-Associated Lymphoproliferative Disorders. | From first dose until first documented progression or death (assessed at 24 months)
  Proportion of patients without disease progression at 24 months per Lugano 2014 criteria.

IPD SHARING:
Plan to Share IPD: No